CLINICAL TRIAL: NCT00000478
Title: Asymptomatic Cardiac Ischemia Pilot (ACIP) Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 67
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2002-02

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia | interventions — Atenolol; Nifedipine; Diltiazem; Isosorbide Dinitrate; Coronary Artery Bypass; Angioplasty, Balloon, Coronary

INTERVENTIONS:
Drug: atenolol
Drug: nifedipine
Drug: diltiazem
Drug: isosorbide dinitrate
Procedure: coronary artery bypass coronary artery bypass
Procedure: angioplasty, transluminal, percutaneous coronary

SUMMARY:
To assess the feasibility of and test the methodology for a full-scale clinical trial of therapies for asymptomatic cardiac ischemia.

DETAILED DESCRIPTION:
BACKGROUND:

Asymptomatic cardiac ischemia, frequently designated as silent myocardial ischemia, refers to episodes of objectively demonstrable transient ischemia in the absence of symptoms. Annually, more than one million patients suffer acute myocardial infarction. Of the approximately 700,000 who are discharged alive from the hospital, as many as 180,000 will be asymptomatic but have evidence of myocardial ischemia on a pre-discharge exercise test. Asymptomatic ischemia has been linked with sudden death or myocardial infarction. It is estimated that in the United States over six million patients have chronic, symptomatic coronary heart disease and up to three million of these may exhibit transient asymptomatic myocardial ischemia. Asymptomatic ischemia is thought to be present in the majority of coronary heart disease patients with stable angina pectoris, over 70 percent of all ischemic episodes being asymptomatic. Asymptomatic ischemia following myocardial infarction or in the presence of chronic stable angina may be associated with substantially increased morbidity and mortality

Traditionally, treatment of patients with coronary heart disease has been given for and guided by patients' symptoms. There was a growing trend toward recognizing asymptomatic cardiac ischemia and according it importance equal to that of symptomatic ischemia. Many physicians believed that suppression of asymptomatic ischemia in patients with coronary heart disease would reduce morbidity and mortality. This was leading to rapidly increasing and widespread applications of both medical and revascularization therapies.

In 1989, there was a lack of knowledge as to the relative efficacy of different treatment strategies to control asymptomatic cardiac ischemia. Given the estimated high prevalence of asymptomatic cardiac ischemia in patients with coronary heart disease and evidence of increased risk of untoward outcome, the public health problem was of sufficient magnitude to warrant a pilot study to determine to what extent asymptomatic ischemia could be controlled. If the pilot study demonstrated feasibility, a full-scale clinical trial would then be considered to evaluate the impact of effective treatment of asymptomatic ischemia on survival and cardiovascular morbidity in patients with coronary heart disease.

DESIGN NARRATIVE:

A total of 1,959 patients were screened by AECG monitoring; 49 percent had asymptomatic ischemia, and 65 percent were enrolled in the study. The 618 patients were randomized to one of the three treatment strategies: 202 to angina-guided medical strategy with titration of anti-ischemic medication to relieve angina; 202 to angina-guided plus AECG ischemia-guided medical strategy with titration of anti-ischemic medication to eliminate both angina and AECG ischemia; and 212 to revascularization by angioplasty or bypass surgery. Patients able to take either beta-adrenergic blocking agents or calcium antagonists were also randomized to receive one of two medical combination regimens: atenolol plus nifedipine or diltiazem plus isosorbide dinitrate. Those who could be treated with only one regimen, such as asthmatic patients, were assigned to the appropriate regimen. The primary outcome was the absence of ischemia at twelve weeks. Recruitment ended in January 1993. Clinical based follow-up was completed for 18 months and survival status free of MI was completed for 24 months

ELIGIBILITY:
Men aand women with angiographically documented coronary artery disease, ischemia on both stress (exercise) testing and 48-hour ambulatory electrocardiogram monitoring, and who were amenable to revascularization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1990-11; Study Completion 1997-06

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Cohen — St. Louis University; Richard Davies — University of Ottawa; John Deanfield — St. Bartholomew's Hospital, University of London; Mark Ketterer — Henry Ford Hospital; Genell Knatterud; Hiltrud Mueller — Montefiore Medical Center; Pamela Ouyang — Johns Hopkins University; Carl Pepine — University of Florida; Craig Pratt — Baylor College of Medicine; William Rogers — University of Alabama at Birmingham; Andrew Selwyn — Brigham and Women's Hospital

REFERENCES:
- [Background] Pepine CJ, Geller NL, Knatterud GL, Bourassa MG, Chaitman BR, Davies RF, Day P, Deanfield JE, Goldberg AD, McMahon RP, et al. The Asymptomatic Cardiac Ischemia Pilot (ACIP) study: design of a randomized clinical trial, baseline data and implications for a long-term outcome trial. J Am Coll Cardiol. 1994 Jul;24(1):1-10. doi: 10.1016/0735-1097(94)90534-7. PMID 8006249
- [Background] Knatterud GL, Bourassa MG, Pepine CJ, Geller NL, Sopko G, Chaitman BR, Pratt C, Stone PH, Davies RF, Rogers WJ, et al. Effects of treatment strategies to suppress ischemia in patients with coronary artery disease: 12-week results of the Asymptomatic Cardiac Ischemia Pilot (ACIP) study. J Am Coll Cardiol. 1994 Jul;24(1):11-20. doi: 10.1016/0735-1097(94)90535-5. PMID 8006252
- [Background] Deedwania PC. Is there evidence in support of the ischemia suppression hypothesis? J Am Coll Cardiol. 1994 Jul;24(1):21-4. doi: 10.1016/0735-1097(94)90536-3. No abstract available. PMID 8006267
- [Background] McMahon RP, Proschan M, Geller NL, Stone PH, Sopko G. Sample size calculation for clinical trials in which entry criteria and outcomes are counts of events. ACIP Investigators. Asymptomatic Cardiac Ischemia Pilot. Stat Med. 1994 Apr 30;13(8):859-70. doi: 10.1002/sim.4780130806. PMID 8047740
- [Background] Tamesis B, Stelken A, Byers S, Shaw L, Younis L, Miller DD, Chaitman BR. Comparison of the Asymptomatic Cardiac Ischemia Pilot and modified Asymptomatic Cardiac Ischemia Pilot versus Bruce and Cornell exercise protocols. Am J Cardiol. 1993 Sep 15;72(9):715-20. doi: 10.1016/0002-9149(93)90891-f. PMID 8249851
- [Background] Chaitman BR, Stone PH, Knatterud GL, Forman SA, Sopko G, Bourassa MG, Pratt C, Rogers WJ, Pepine CJ, Conti CR. Asymptomatic Cardiac Ischemia Pilot (ACIP) study: impact of anti-ischemia therapy on 12-week rest electrocardiogram and exercise test outcomes. The ACIP Investigators. J Am Coll Cardiol. 1995 Sep;26(3):585-93. doi: 10.1016/0735-1097(95)00013-t. PMID 7642847
- [Background] Bourassa MG, Pepine CJ, Forman SA, Rogers WJ, Dyrda I, Stone PH, Chaitman BR, Sharaf B, Mahmarian J, Davies RF, et al. Asymptomatic Cardiac Ischemia Pilot (ACIP) study: effects of coronary angioplasty and coronary artery bypass graft surgery on recurrent angina and ischemia. The ACIP investigators. J Am Coll Cardiol. 1995 Sep;26(3):606-14. doi: 10.1016/0735-1097(95)00005-o. PMID 7642849
- [Background] Conti RC, Kantterud GL, Sopko G: Correction. Letter to Editor. J Am Coll Cardiol 26:842, 1995
- [Background] Caracciolo EA, Chaitman BR, Forman SA, Stone PH, Bourassa MG, Sopko G, Geller NL, Conti CR. Diabetics with coronary disease have a prevalence of asymptomatic ischemia during exercise treadmill testing and ambulatory ischemia monitoring similar to that of nondiabetic patients. An ACIP database study. ACIP Investigators. Asymptomatic Cardiac Ischemia Pilot Investigators. Circulation. 1996 Jun 15;93(12):2097-105. doi: 10.1161/01.cir.93.12.2097. PMID 8925577
- [Background] Bourassa MG, Knatterud GL, Pepine CJ, Sopko G, Rogers WJ, Geller NL, Dyrda I, Forman SA, Chaitman BR, Sharaf B, et al. Asymptomatic Cardiac Ischemia Pilot (ACIP) Study. Improvement of cardiac ischemia at 1 year after PTCA and CABG. Circulation. 1995 Nov 1;92(9 Suppl):II1-7. doi: 10.1161/01.cir.92.9.1. PMID 7586390
- [Background] Pratt CM, McMahon RP, Goldstein S, Pepine CJ, Andrews TC, Dyrda I, Frishman WH, Geller NL, Hill JA, Morgan NA, Stone PH, Knatterud GL, Sopko G, Conti CR. Comparison of subgroups assigned to medical regimens used to suppress cardiac ischemia (the Asymptomatic Cardiac Ischemia Pilot [ACIP] Study). Am J Cardiol. 1996 Jun 15;77(15):1302-9. doi: 10.1016/s0002-9149(96)00196-8. PMID 8677870
- [Background] Pepine CJ, Andrews T, Deanfield JE, Forman S, Geller N, Hill JA, Pratt C, Rogers WJ, Sopko G, Steingart R, Stone PH, Conti CR. Relation of patient characteristics to cardiac ischemia during daily life activity (an Asymptomatic Cardiac Ischemia Pilot Data Bank Study). Am J Cardiol. 1996 Jun 15;77(15):1267-72. doi: 10.1016/s0002-9149(96)00190-7. PMID 8677864
- [Background] Conti CR, Bourassa MG, Chaitman BR, Geller NL, Knatterud GL, Pepine CJ, Pratt C, Sopko G. Asymptomatic cardiac ischemia pilot (ACIP). Trans Am Clin Climatol Assoc. 1995;106:77-83; discussion 83-4. PMID 7483181
- [Background] Stone PH, Chaitman BR, McMahon RP, Andrews TC, MacCallum G, Sharaf B, Frishman W, Deanfield JE, Sopko G, Pratt C, Goldberg AD, Rogers WJ, Hill J, Proschan M, Pepine CJ, Bourassa MG, Conti CR. Asymptomatic Cardiac Ischemia Pilot (ACIP) Study. Relationship between exercise-induced and ambulatory ischemia in patients with stable coronary disease. Circulation. 1996 Oct 1;94(7):1537-44. doi: 10.1161/01.cir.94.7.1537. PMID 8840841
- [Background] Sharaf BL, Williams DO, Miele NJ, McMahon RP, Stone PH, Bjerregaard P, Davies R, Goldberg AD, Parks M, Pepine CJ, Sopko G, Conti CR. A detailed angiographic analysis of patients with ambulatory electrocardiographic ischemia: results from the Asymptomatic Cardiac Ischemia Pilot (ACIP) study angiographic core laboratory. J Am Coll Cardiol. 1997 Jan;29(1):78-84. doi: 10.1016/s0735-1097(96)00444-5. PMID 8996298
- [Background] Davies RF, Goldberg AD, Forman S, Pepine CJ, Knatterud GL, Geller N, Sopko G, Pratt C, Deanfield J, Conti CR. Asymptomatic Cardiac Ischemia Pilot (ACIP) study two-year follow-up: outcomes of patients randomized to initial strategies of medical therapy versus revascularization. Circulation. 1997 Apr 15;95(8):2037-43. doi: 10.1161/01.cir.95.8.2037. PMID 9133513
- [Background] Conti CR, Geller NL, Knatterud GL, Forman SA, Pratt CM, Pepine CJ, Sopko G. Anginal status and prediction of cardiac events in patients enrolled in the asymptomatic cardiac ischemia pilot (ACIP) study. ACIP investigators. Am J Cardiol. 1997 Apr 1;79(7):889-92. doi: 10.1016/s0002-9149(97)00009-x. PMID 9104900
- [Background] Pepine CJ, Sharaf B, Andrews TC, Forman S, Geller N, Knatterud G, Mahmarian J, Ouyang P, Rogers WJ, Sopko G, Steingart R, Stone PH, Conti CR. Relation between clinical, angiographic and ischemic findings at baseline and ischemia-related adverse outcomes at 1 year in the Asymptomatic Cardiac Ischemia Pilot study. ACIP Study Group. J Am Coll Cardiol. 1997 Jun;29(7):1483-9. doi: 10.1016/s0735-1097(97)00083-1. PMID 9180108
- [Background] Steingart RM, Forman S, Coglianese M, Bittner V, Mueller H, Frishman W, Handberg E, Gambino A, Knatterud G, Conti CR. Factors limiting the enrollment of women in a randomized coronary artery disease trial. The Asymptomatic Cardiac Ischemia Pilot Study (ACIP) Investigators. Clin Cardiol. 1996 Aug;19(8):614-8. doi: 10.1002/clc.4960190807. PMID 8864334
- [Background] Stone PH, Chaitman BR, Forman S, Andrews TC, Bittner V, Bourassa MG, Davies RF, Deanfield JE, Frishman W, Goldberg AD, MacCallum G, Ouyang P, Pepine CJ, Pratt CM, Sharaf B, Steingart R, Knatterud GL, Sopko G, Conti CR. Prognostic significance of myocardial ischemia detected by ambulatory electrocardiography, exercise treadmill testing, and electrocardiogram at rest to predict cardiac events by one year (the Asymptomatic Cardiac Ischemia Pilot [ACIP] study). Am J Cardiol. 1997 Dec 1;80(11):1395-401. doi: 10.1016/s0002-9149(97)00706-6. PMID 9399710
- [Background] Mahmarian JJ, Steingart RM, Forman S, Sharaf BL, Coglianese ME, Miller DD, Pepine CJ, Goldberg AD, Bloom MF, Byers S, Dvorak L, Pratt CM. Relation between ambulatory electrocardiographic monitoring and myocardial perfusion imaging to detect coronary artery disease and myocardial ischemia: an ACIP ancillary study. The Asymptomatic Cardiac Ischemia Pilot (ACIP) Investigators. J Am Coll Cardiol. 1997 Mar 15;29(4):764-9. doi: 10.1016/s0735-1097(96)00572-4. PMID 9091522
- [Background] Rogers WJ, Bourassa MG, Andrews TC, Bertolet BD, Blumenthal RS, Chaitman BR, Forman SA, Geller NL, Goldberg AD, Habib GB, et al. Asymptomatic Cardiac Ischemia Pilot (ACIP) study: outcome at 1 year for patients with asymptomatic cardiac ischemia randomized to medical therapy or revascularization. The ACIP Investigators. J Am Coll Cardiol. 1995 Sep;26(3):594-605. doi: 10.1016/0735-1097(95)00228-v. PMID 7642848
- [Background] Pepine CJ, Bourassa MG, Chaitman BR, Davies RF, Kerensky RA, Sharaf B, Knatterud GL, Forman SA, Pratt CM, Staples ED, Sopko G, Conti CR. Factors influencing clinical outcomes after revascularization in the asymptomatic cardiac ischemia pilot (ACIP). ACIP Study Group. J Card Surg. 1999 Jan-Feb;14(1):1-8. doi: 10.1111/j.1540-8191.1999.tb00943.x. PMID 10678439
- [Background] Pepine CJ, Mark DB, Bourassa MG, Chaitman BR, Davies RF, Knatterud GL, Forman S, Pratt CM, Sopko G, Conti CR. Cost estimates for treatment of cardiac ischemia (from the Asymptomatic Cardiac Ischemia Pilot [ACIP] study). Am J Cardiol. 1999 Dec 1;84(11):1311-6. doi: 10.1016/s0002-9149(99)00563-9. PMID 10614796
- [Background] Frishman WH, Gomberg-Maitland M, Hirsch H, Catanese J, Furia-Palazzo S, Mueller H, Steingart R, Forman S. Differences between male and female patients with regard to baseline demographics and clinical outcomes in the Asymptomatic Cardiac Ischemia Pilot (ACIP) Trial. Clin Cardiol. 1998 Mar;21(3):184-90. doi: 10.1002/clc.4960210310. PMID 9541762
- [Background] Handberg-Thurmond E, Baker A, Coglianese ME, Forman S, Pepine CJ, Geller N, Chaitman B. Identifying high yield sources of patients with coronary artery disease for clinical trials: lessons from the Asymptomatic Cardiac Ischemia Pilot (ACIP) experience. The ACIP Study Group. Clin Cardiol. 1998 Mar;21(3):177-82. doi: 10.1002/clc.4960210308. PMID 9541761
- [Background] Davies RF. The need for a prognosis trial of revascularization and aggressive medical therapy in patients with asymptomatic cardiac ischemia. ACIP Investigators. Asymptomatic Cardiac Ischemia Pilot. Clin Cardiol. 1998 Mar;21(3):154-6. doi: 10.1002/clc.4960210303. No abstract available. PMID 9541757
- [Background] Sharaf BL, Bourassa MG, McMahon RP, Pepine CJ, Chaitman BR, Williams DO, Davies RF, Proschan M, Conti CR. Clinical and detailed angiographic findings in patients with ambulatory electrocardiographic ischemia without critical coronary narrowing: results from the Asymptomatic Cardiac Ischemia Pilot (ACIP) Study. Clin Cardiol. 1998 Feb;21(2):86-92. doi: 10.1002/clc.4960210205. PMID 9491946
- [Background] Asymptomatic Cardiac Ischemia Pilot study (ACIP). Am J Cardiol. 1992 Sep 15;70(7):744-7. doi: 10.1016/0002-9149(92)90552-a. PMID 1519524
- Available data/document: Individual Participant Data Set: ACIP — http://biolincc.nhlbi.nih.gov/studies/acip — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.